CLINICAL TRIAL: NCT03875456
Title: Needle Aspiration for Large Cephalohematoma : a Retrospective Study of Complications
Brief Title: Needle Aspiration for Large Cephalohematoma
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0107
Record Dates: First submitted 2019-03-13; First posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Cephalohematoma
Keywords: Cephalohematoma; Infant, Newborn; Perinatal Care; Plagiocephaly; Nonsynostotic; Skull/pathology
MeSH Terms: conditions — Plagiocephaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The cephalohematoma is a common pathology of newborns. Observation is the primary treatment for the most of small uncomplicated cephalohematoma. However large cephalohematoma can lead to calcification with anesthetic local deformation or deformational plagiocephaly. The objective of the study was to evaluate the iatrogenic risk associated with early puncture on local anesthesia.

DETAILED DESCRIPTION:
This is a retrospective study of 67 newborns followed at the University Hospital of Montpellier between 2010 and 2017. Treatment was puncture under local anesthesia between 2 and 4 weeks of life.

Any potential complication events were searched retrospectively during the month after the puncture. Analyze of the electronic medical record was made as followed: read of peri-operative and post-operative reports, looking for readmission in Pediatric Emergency department and finally read of the report of the clinical control 1 month after the procedure

ELIGIBILITY:
Inclusion criteria:

* diagnosis of cephalohematoma was performed by the two senior plastic pediatric surgeon of the study
* the diagnosis was confirmed by ultrasound examination

Exclusion criteria:

* Skull fracture (seen by ultrasound examination)
* Intra-cranial complication (ultrasound examination)

Ages: 15 Days to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients presenting cephalohematoma
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Complication events during the month after the puncture. | 1 day
  retrospective data collection. Analyze of the electronic medical record was made as followed: read of peri-operative and post-operative reports, looking for readmission in Pediatric Emergency department and finally read of the report of the clinical control 1 month after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume CAPTIER, MD.PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France